CLINICAL TRIAL: NCT00531271
Title: A Phase I/II Trial of ABI-008 (Nab-docetaxel) in Patients With Metastatic Breast Cancer
Brief Title: ABI-008 Trial in Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA302
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABI-008 (nab-docetaxel) — ABI-008; 60-200 mg/m²; Intravenous infusion every 3 weeks.

SUMMARY:
To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of ABI-008 giver every 3 weeks; to characterize the toxicities of ABI-008; and to determine the pharmacokinetic parameters for ABI-008 when given on an every-3-week schedule to patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

Phase I Study

Each subject must meet the following criteria to be enrolled in this study.

1. Pathologically confirmed adenocarcinoma of the breast with metastasis.
2. No more than 2 prior chemotherapy regimen for metastatic breast cancer. Patient should have received anthracycline and may have received a taxane but not within 6 months for registration on the study.
3. Patient may have measurable or evaluable disease.
4. Patient may have non-measurable bone only disease.
5. At least 4 weeks since prior cytotoxic chemotherapy. Patients should have recovered from all acute effects of such therapy.
6. At least 4 weeks since radiotherapy, with full recovery.
7. At least 4 weeks since recovery from major surgery, with full recovery.
8. ECOG performance status 0-2.
9. Age ≥18 years.
10. Patient must have the following blood counts at Baseline:

    * WBC > 3.0 x 109 cells/L;
    * ANC ≥ 1.5 x 109 cells/L;
    * Platelets ≥ 100 x 109 cells/L;
    * Hgb ≥ 9 grams/dL.
11. Patient has the following blood chemistry levels at Baseline:

    * AST (SGOT), ALT (SGPT) ≤ 1.5x upper limit of normal range (ULN);
    * Total Bilirubin < ULN;
    * Alkaline phosphatase ≤ 2.5x ULN (unless bone metastasis is present in the absence of liver metastasis);
    * Creatinine ≤ 1.5 mg/dL.
12. Peripheral neuropathy Grade 0 or stable Grade 1, by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0.
13. If female of childbearing potential, serum pregnancy test is negative (within 72 hours of the first dose of study drug).
14. If fertile, the patient agrees to use an effective method to avoid pregnancy for the duration of the study.
15. Life expectancy should be ≥ 3 months.
16. Informed consent document has been obtained stating that the patient understands the investigational nature of the proposed treatment.
17. If obese, a patient must be treated with doses calculated using his/her actual body surface area (BSA) (the physician must be comfortable treating at the full BSA dose regardless of BSA).

Phase II Study

1. Pathologically confirmed adenocarcinoma of the breast with metastasis.
2. Patients should have not received prior chemotherapy for their metastatic disease. If a taxane is used as adjuvant or neoadjuvant therapy, at least 12 months should have elapsed from the date of the last dose.
3. Patient must have at least one measurable metastatic lesion.
4. At least 4 weeks since prior cytotoxic chemotherapy. Patients should have recovered from all acute effects of such therapy.
5. At least 4 weeks since radiotherapy, with full recovery.
6. At least 4 weeks since major surgery, with full recovery.
7. ECOG performance status 0-2.
8. Age ≥18 years.
9. Patient must have the following blood counts at Baseline:

   * WBC > 3.0 x 109 cells/L;
   * ANC ≥ 1.5 x 109 cells/L;
   * Platelets ≥ 100 x 109 cells/L;
   * Hgb ≥ 9 grams/dL.
10. Patient has the following blood chemistry levels at Baseline:

    * AST (SGOT), ALT (SGPT) ≤ 1.5x upper limit of normal range (ULN);
    * Total Bilirubin < ULN;
    * Alkaline phosphatase ≤ 2.5x ULN (unless bone metastasis is present in the absence of liver metastasis);
    * Creatinine ≤ 1.5 mg/dL.
11. Peripheral neuropathy Grade 0 or stable Grade 1, by NCI CTCAE v3.0.
12. If female of childbearing potential, serum pregnancy test is negative (within 72 hours of the first dose of study drug).
13. If fertile, the patient agrees to use an effective method to avoid pregnancy for the duration of the study.
14. Life expectancy should be ≥ 3 months.
15. Informed consent document has been obtained stating that the patient understands the investigational nature of the proposed treatment.

Exclusion Criteria:

Phase I Study

Subjects who meet any of the following criteria will be excluded from the study.

1. Concurrent therapy (chemotherapy, hormonal therapy, kinase inhibitors, immunotherapy, etc) for breast cancer. Bisphosphonates are allowed.
2. Parenchymal brain metastases, unless documented to be clinically and radiographically stable for at least 6 months after treatment.
3. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Patients with significant cardiovascular disease including congestive heart failure (New York Heart Association Class III or IV), active angina pectoris or recent myocardial infarction (within the last 6 months).
5. History of other malignancy within the last 5 years which could affect the diagnosis or assessment of breast cancer excluding non-melanomatous skin cancer and cervical carcinoma in situ.
6. Patients who have received an investigational drug within the previous 4 weeks.
7. Patient is currently enrolled in any other clinical study in which investigational procedures are performed or investigational therapies are administered. A patient may not enroll in such clinical trials while participating in this study.
8. Pregnant or nursing women.
9. Patients with history of allergic reactions attributed to solvent-based docetaxel(Taxotere).
10. ECOG performance status 3-4.
11. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with docetaxel. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.

Phase II Study

Subjects who meet any of the following criteria will be excluded from the study.

1. Prior neo-adjuvant or adjuvant chemotherapy is allowed. If a taxane was part of the adjuvant regimen, at least 12 months should have transpired since completion of taxane regimen.
2. Concurrent therapy (chemotherapy, hormonal therapy, kinase inhibitors, immunotherapy, etc) for breast cancer.
3. Parenchymal brain metastases, unless documented to be clinically and radiographically stable for at least 6 months after treatment.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
5. Patients with significant cardiovascular disease including congestive heart failure (New York Heart Association Class III or IV), active angina pectoris or recent myocardial infarction (within the last 6 months).
6. History of other malignancy within the last 5 years which could affect the diagnosis or assessment of breast cancer excluding non-melanomatous skin cancer and cervical carcinoma in situ.
7. Patients who have received an investigational drug within the previous 4weeks.
8. Patient is currently enrolled in any other clinical study in which investigational procedures are performed or investigational therapies are administered.
9. Pregnant or nursing women.
10. Patients with history of allergic reactions attributed to solvent-based docetaxel(Taxotere).
11. ECOG performance status 3-4.
12. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with docetaxel.
13. Patients with tumor overexpression of HER2/neu.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2007-11-01 (Actual); Primary Completion 2008-12-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose limiting toxicities (DLTs) of ABI-008 giver every three weeks. | End of Study (EOS) and Follow Up

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of ABI-008 in the metastatic breast cancer patient population; and to determine the pharmacokinetic parameters for ABI-008 when given on an every-3-week schedule. | End of Study (EOS) and Follow Up

CONTACTS AND LOCATIONS:
Overall Officials: Nuhad Ibrahim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States